CLINICAL TRIAL: NCT02507895
Title: Brain-Computer Interface-Assisted Motor Imagery for Gait Retraining in Neurorehabilitation
Brief Title: Effect of Brain-Computer Interfaced-Assisted Motor Imagery for Gait Retraining in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University Health System, Singapore (Other); Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCI-LL2012/00658
Record Dates: First submitted 2014-12-21; First posted 2015-07-24 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2017-11

CONDITIONS: Stroke
Keywords: Stroke; lower extremeties; Brain-computer interface; Motor imagery; Rehabilitation; TMS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MI-BCI training (Experimental): subjects will undergo 12 sessions over 4 weeks of MI-BCI training
  Interventions: Device: MI-BCI

INTERVENTIONS:
Device: MI-BCI — Subjects will be seated comfortably in front of a computer screen. An EEG cap will be comfortably worn over the head of the subject to record EEG traces of any activated cortical areas. If subjects are able to activate the device and are agreeable to participate in the second phase of the study, they will be enrolled in a 4-week BCI-MI training program of 12 sessions. Subjects will be required to perform 160 trials of MI altogether with assigned rest periods (5 mins) every 40 trials. Each session will last approximate 45 minutes excluding set up time.

SUMMARY:
Currently the process for stroke recovery is slow with majority of its treatments focused around physical therapy. Among the many methods employed to facilitate recovery in stroke, the use of motor imagery (MI) training may be beneficial towards stroke rehabilitation.

In the current study, we propose 2 aims. Our first aim is to determine the feasibility and efficacy of a novel brain-computer interface-assisted MI train program (BCI-MI) in patients with chronic ischemic stroke. This is designed as a proof-of-concept study that only require a single-session trial. If patients successfully activate the BCI-MI system without much difficulty, our second aim is to enroll patients into a 4-week training program using the BCI-MI. Both functional magnetic resonance imaging (fMRI) and transcranial magnetic stimulation (TMS) will be done to determine the effects of the 4-week training program. Subjects may potentially see improvements in walking gait as preliminary data from previous studies have demonstrated positive results.

DETAILED DESCRIPTION:
In the first study, we propose 20 subjects who have sustained their first ever haemorrhagic or ischaemic subcortical stroke with lower limb impairment more than 9 months prior to study enrollment. Subjects will be recruited from the existing patients on the study physician's cohort of patients and from referrals from attending physicians. During the initial screening visit, it will be ascertained that subject fulfills criteria for participation and informed consent will be obtained by study staff. Subjects will be fully briefed in detail regarding the experimental procedure, risk and benefits involved and their responsibilities during the study.

Once consent is provided, subjects will undergo a MI-BCI usability session, they will be seated comfortably in front of a computer screen. An EEG cap will be comfortably worn over the head of the subject to record EEG traces of any activated cortical areas. Subjects will then be instructed to perform a mental imagery task whereby they will imagine themselves walking properly with their affected leg. The accuracies in classifying correct motor imagery from the idle condition from EEG will be recorded for each subject. Subjects who obtain an accuracy of more than 57.5% are considered eligible for the MI-BCI training program. Subjects eligible for the MI-BCI training will then undergo a series of functional assessments, including (1) functional clinical measures (10 meter walk test and Up-to-Go test), (2) gait analysis , (3) cortical activity assessment using TMS, and (4) MRI and DTI scan. (5) Psychological tests including Beck Depression Inventory, fatigue severity scale, digital span test. Before the start of MI-BCI training, subjects will undergo one more MI-BCI session of calibration, which will be performed totally the same with BCI usability session to gather more valuable data for analyzing. After finishing all 5 assessments and MI-BCI calibration session, the MI-BCI training can be started at the frequency of 3 times a week lasting for 4 weeks. The procedure of MI-BCI training is identical to the one in BCI usability session except that a cartoon character in the computer screen will be activated to walk forward if subjects successfully perform an accurate mental imagery. Subjects undergoing MI-BCI training will be required to perform 160 trials of MI altogether with assigned rest periods (5 mins) every 40 trials. Each session will last approximate 45 minutes excluding set-up time. The number of times subjects can successfully perform the MI task and the ease in which they are able to perform the task will be recorded. Distinct brain signals such as event-related desynchronization or synchronization (ERD/ERS) are detectable on EEG for both real and imagined motor movements in healthy subjects. Using this technique, MI-BCI, which translates the imagination of movements into online commands, provides a promising neural communication system for stroke patients who suffer from motor disabilities. We have previously collaborated with I2R-A*STAR BCI to design a custom-built BCI software to sync with an EEG amplifier. We have demonstrated the efficacy of this custom-built MI-BCI device on upper limb stroke impairments, therefore, the procedure and equipment used will be kept identical except for the software interface, which shows a cartoon character on the screen. Subjects will undergo the same five assessments again at the end of the 4-week's MI-BCI training and 4-6 weeks after the last session of MI-BCI training, respectively, including (1) functional clinical outcome measures (10 meter walk test and Up-to-Go test), (2) gait analysis, (3) cortical activity assessment using TMS, and (4) MRI and DTI. (5) Psychological tests including Beck Depression Inventory, fatigue severity scale, digital span test.

The timed up-and-go test is a measurement of mobility. It includes a number of tasks such as standing from a seating position, walking, turning, stopping, and sitting down. For the test, the person is asked to stand up from a standard chair and walk a distance of approximately 3 meters, turn around and walk back to the chair and sit down again. The 10 meter walk test is a test of walking speed. Timed up-to-go test and 10 meter walk test will be assessed by certified physical therapist or trained research staff, and will take approximate 30 minutes including set-up time.

Gait analysis is the systematic study of locomotion. It will be performed in NUH, by a certified medical technician or a trained research staff. Subjects will be required to wear shorts and the whole trial process might be video-recorded for future analyzing the quality of subjects' movement (face will not be captured and consent will be obtained in advance). Markers might be worn at various points of reference of the body such as iliac spines of the pelvis, ankle malleolus, and the condyles of the knee. Electromyography (EMG) sensors might be worn at the area of quadriceps femoris,hamstring, gastrocnemius and tibialis anterior muscles for both legs. Gait parameters of temporal and spatial measures and joint kinematics will be recorded while the subject is walking along the walkway with a force platform, according to the instruction of the medical technician or the trained research staff. Each session will last approximate 1 hour including set-up time.

TMS will be performed to investigate the mechanisms of this training on cortical plasticity as indexed by cortical excitability changes. For the MEP study, we will initially adjust TMS intensity to achieve a baseline MEP in the tibialis anterior muscle of the leg to about 1 mV peak-to-peak amplitude before intervention. Stimulation intensity will be kept constant for each subject throughout the study. The MEPs will be recorded in a computer for off-line analysis. We will record 10 MEPs for each time and average their peak-to-peak amplitude. For the paired pulse stimulation, a first subthreshold conditioning stimulus will be applied, followed at a variable interstimulus interval (ISI), by a second suprathreshold stimulus. We will use the following ISIs - 2, 3, 4, 6, 9, 10, 12, 15 ms. The percentage of change for each ISI before and after treatment will be calculated from the MEPs and will therefore important to measure changes in intracortical facilitation and inhibition. Each session will last approximate 1 hour including set-up time.

MRI/DTI scan will be performed at CIRC, NUS. Prior to the scan, all patients will be briefed of the test procedure and safety aspects. A medically-trained physician will be on standby throughout the procedure. All participants will be scanned on a 3-T GE scanner using a standard radiofrequency head coil. Head motion was minimized by foam padding and forehead-restraining straps. A T1-weighted high-resolution scan and a set of axial fluid attenuated inversion recovery images will be acquired. T1-weighted and fluid attenuated inversion recovery images will be realigned and spatially normalized into images of isotropic voxel size implemented in Matlab. Each session will last approximate 1 hour including set-up time.

A research staff will administer Beck Depression Inventory (BDI), Fatigue Severity Scale (FSS), forward and backward digit span for controlling for confounding effect of cognitive improvement in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 21-70 years;
* first ever haemorrhagic or ischaemic hemiplegic stroke more than 9 months prior to study enrollment;
* Functional Ambulatory Category 3-4 (requires not more than minimal assistance for walking)

Exclusion Criteria:

* Severe claustrophobia;
* pregnancy;
* cardiac pacemakers;
* orthodontics (braces);
* metal implant;
* presence of other non MR-compatible ferromagnetic implants;
* history of epilepsy;
* sensorimotor disturbance due to other causes other than stroke;
* severe pain in the lower limbs affecting gait;
* uncontrolled medical conditions including hypertension, diabetes mellitus and unstable angina;
* major depression and a history of psychotic disorders.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
changes of " gait parameters measured by " from baseline to post-training and 4-6 weeks after training | baseline, 5 min after training, 4-6 weeks after training
  Gait analysis will be performed using the Tekscan walkway system. Subjects will be required to walk on a mat at their comfort speed. Gait parameters including step and stride parameters, symmetry scores, velocity, and cadence temporal will be collected and recorded while the subject is walk along the walkway.

SECONDARY OUTCOMES:
Changes of "cortical excitability measured by TMS" from baseline to post-training and 4-6 weeks after training | baseline, 5 min after training, 4-6 weeks after training
  Motor threshold will be measured according to the technique described by Rossini et al. (1994). For the MEP study, we will initially adjust TMS intensity to achieve a baseline MEP in the tibialis anterior muscle of the leg to about 1 mV peak-to-peak amplitude before intervention. Stimulation intensity will be kept constant for each subject throughout the study. We will record 10 MEPs for each time and average their peak-to-peak amplitude and area under-the-curve. For the paired-pulse stimulation, a first subthreshold conditioning stimulus will be applied, followed at a variable interstimulus interval (ISI), by a second suprathreshold stimulus. We will use the following ISIs - 2, 3, 4, 6, 9, 10, 12, 15 ms. The percentage of change for each ISI before and after treatment will be calculated from the MEPs and will therefore important to measure changes in intracortical facilitation and inhibition. Each session will last approximate 1 hour including set-up time.
changes of " cortical excitability measured by fMRI/DTI" from baseline to post-training and 4-6 weeks after training | baseline, 5 min after training, 4-6 weeks after training
  All subjects will be asked to make their way on their own to CIRC, NUS. The patients are currently treated in an outpatient setting and their condition is stable. A research assistant will be onsite to meet the patient at CIRC and run through the whole procedure with the patient. Prior to the scan, all patients will be briefed of the test procedure and safety aspects. A medically-trained physician will be on standby throughout the procedure. All participants will be scanned on a 3-T GE scanner using a standard radiofrequency head coil. Head motion was minimized by foam padding and forehead-restraining straps. A T1-weighted high-resolution scan and a set of axial fluid attenuated inversion recovery images will be acquired. T1-weighted and fluid-attenuated inversion recovery images will be realigned and spatially normalized into images of isotropic voxel size implemented in Matlab. Each session will last approximate 1 hour including set-up time.
Mobility changes from baseline to post-training and 4-6 weeks after training, as measured by "timed up-and-go test" | baseline, 5 min after training, 4-6 weeks after training
  The timed up-and-go test is a measurement of mobility. It includes a number of tasks such as standing from a seating position, walking, turning, stopping, and sitting down. For the test, the person is asked to stand up from a standard chair and walk a distance of approximately 3 meters, turn around and walk back to the chair and sit down again.
changes of walking speed measured by "10 metre walk test", from baseline to post-training and 4-6 weeks after training | baseline, 5 min after training, 4-6 weeks after training
  The 10 meter walk test is a test of walking speed.

CONTACTS AND LOCATIONS:
Overall Officials: Effie Chew, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Dunsky A, Dickstein R, Ariav C, Deutsch J, Marcovitz E. Motor imagery practice in gait rehabilitation of chronic post-stroke hemiparesis: four case studies. Int J Rehabil Res. 2006 Dec;29(4):351-6. doi: 10.1097/MRR.0b013e328010f559. PMID 17106356
- [Background] Dunsky A, Dickstein R, Marcovitz E, Levy S, Deutsch JE. Home-based motor imagery training for gait rehabilitation of people with chronic poststroke hemiparesis. Arch Phys Med Rehabil. 2008 Aug;89(8):1580-8. doi: 10.1016/j.apmr.2007.12.039. PMID 18674992